CLINICAL TRIAL: NCT02610283
Title: A Randomized, Double-Blind, Placebo Controlled , Phase 2 Study to Evaluate the Efficacy and Safety of QPI-1002 for the Prevention of Acute Kidney Injury in Subjects at High Risk for AKI Following Cardiac Surgery
Brief Title: A Study to Evaluate Efficacy and Safety of QPI-1002 for Prevention of Acute Kidney Injury Following Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Quark Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QRK209
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2018-04

CONDITIONS: Acute Kidney Injury
Keywords: AKI
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QPI-1002 (Active Comparator): QPI-1002 Injection, single dose
  Interventions: Drug: QPI-1002
- Placebo (Placebo Comparator): isotonic saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QPI-1002 — IV injection
  Arms: QPI-1002
Drug: Placebo — isotonic saline
  Arms: Placebo

SUMMARY:
This trial is designed to evaluate QPI-1002 versus placebo for the prevention of AKI in subjects who are at high risk for AKI following cardiac surgery. Half of the participants will receive QPI-1002 while the other half will receive placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, Phase 2 trial to evaluate QPI-1002 versus placebo for the prevention of AKI in subjects who are at high risk for AKI following cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to understand the requirements of the study, are able to provide written informed consent and are willing and able to comply with the requirements of the study
* Male or female, age ≥ 45 years old.
* Have stable renal function per Investigator assessment and no known increase in serum creatinine of ≥ 0.3 mg/dL during preceding 4 weeks.
* Scheduled to undergo non-emergent open chest cavity cardiovascular surgeries, including use of coronary pulmonary bypass (CPB) and no CPB:

  * Combined coronary artery bypass grafting (CABG) surgery and surgery of one or more cardiac valve (valve(s) surgery) and at least 1 AKI Risk Factor;
  * Surgery of more than one cardiac valve (valve surgery) and at least 1 AKI Risk Factor;
  * Surgery of the aortic root or ascending part of the aorta, or in combination with the aortic valve, and at least 1 AKI Risk Factor; circulatory arrest is not excluded;
  * Aortic root or ascending part of the aorta, combined with CABG and/or valve(s) surgery and at least 1 AKI Risk Factor; circulatory arrest is not excluded;
  * If only CABG or single valve surgery, subjects are required to have at least 2 AKI Risk Factors:

AKI Risk Factors:

* Age ≥ 70 years
* eGFR ≤ 60 ml/min/1.73m2 by CKD-EPI formula at Screening.
* Diabetes (Type 1 or 2), requiring at least 1 oral hypoglycemic agent or insulin
* Proteinuria ≥ 0.3g/d, spot UPCR ≥ 0.3g/gm or urine dip stick ≥ +2
* History of congestive heart failure requiring hospitalization

Exclusion Criteria:

* Have an eGFR ≤ 20 mL/min/1.73 m2
* Subjects with an eGFR ≤ 60 mL/min/1.73 m2 requiring intravascular iodinated contrast within 48 hours of the day of surgery. However, subjects may be included if the post contrast increase in serum creatinine is < 0.3 mg/dl in at least 2 serum creatinine evaluations performed not less than 36 hours apart.
* Have a history of any organ or cellular transplant which requires active immunosuppressive treatment which can interfere with kidney function
* Emergent surgeries, including aortic dissection, and major congenital heart defects
* Scheduled to undergo transcatheter aortic valve implantation (TAVI) or transcatheter aortic valve replacement (TAVR) or single vessel, mid-CAB off-pump surgeries or left ventricular assist device (LVAD) implantation
* Have participated in an investigational drug study in the last 30 days
* Have a known allergy to or had participated in a prior study with siRNA
* Have a history of human immunodeficiency virus (HIV) infection
* Have known active Hepatitis B (HBV) (Note: Subjects with a serological profile suggestive of clearance, or prior antiviral treatment of HBV infection may be enrolled)
* Are HCV-positive (detectable HCV RNA) (Note: Subjects at least 24 weeks from completion of treatment with an antiviral regimen and who remain free of HCV as determined by HCV RNA testing may be enrolled.)
* Have had cardiogenic shock or hemodynamic instability within the 24 hours prior to surgery, requiring inotropes or vasopressors or other mechanical devices such as intra-aortic balloon counter-pulsation (IABP)
* Have required any of the following within a week prior to cardiac surgery: defibrillator or permanent pacemaker, mechanical ventilation, IABP, left ventricular assist device (LVAD), other forms of mechanical circulatory support (MCS) (Note: The prophylactic insertion of an IABP preoperatively for reasons not related to existing LV pump function is not exclusionary).
* Have required cardiopulmonary resuscitation within 14 days prior to cardiac surgery
* Have ongoing sepsis or history of sepsis within the past 2 weeks or untreated diagnosed infection prior to Screening visit. Sepsis is defined as presence of a confirmed pathogen, along with fever or hypothermia, and hypoperfusion or hypotension
* Have total bilirubin or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the upper limit of normal (ULN) at time of screening
* Have Child Pugh Class A liver disease with ALT/AST above the upper limit of normal or Class B or higher. (This criterion is only applicable in a patient population with underlying chronic liver disease, i.e., cirrhosis.)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2015-12; Primary Completion 2018-02 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects developing AKI as defined by the AKIN criteria | Baseline through Day 5

SECONDARY OUTCOMES:
Proportion of subjects developing at least on of the following events: death, needing renal replacement therapy (RRT) during the 90-day post-operative period, or having a ≥ 25% reduction in SCr based eGFR at the Day 90 visit | Baseline through Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Squiers, M.D., Study Director — Quark Pharmaceuticals
Locations (36):
- United States (20):
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - University of Florida, Gainesville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - River City Clinical Research, Jacksonville, Florida
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Indiana Ohio Heart, Fort Wayne, Indiana
  - St. Vincent Medical Group, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Mid Michigan Cardiovascular Research, Midland, Michigan
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Washington University, St Louis, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Lindner Research Center, The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Baylor University, Dallas, Texas
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (8):
  - St. John Regional Hospital, Saint John, New Brunswick
  - Hamilton Health Sciences, Hamilton, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Centre hospitalier de l'universite de Montreal, Montreal, Quebec
  - Mcgill University Health Center - Royal Victoria Hospital, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Instiut Universitaire de Cardiologie et Pneumologie de Quebec, Québec, Quebec
- Germany (8):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinikum der Universität zu Köln, Cologne
  - Herzzentrum Dresden GmbH, Dresden
  - Westdeutsches Herzzentrum Essen / Universitätsklinikum Essen, Essen
  - Universitätsklinikum Giessen und Marburg / Standort Giessen / Zentrum für Chirurgie, Giessen
  - Universitätsklinikum Heidelberg, Heidelberg
  - Herzzentrum Leipzig GmbH, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz

REFERENCES:
- [Derived] Thielmann M, Corteville D, Szabo G, Swaminathan M, Lamy A, Lehner LJ, Brown CD, Noiseux N, Atta MG, Squiers EC, Erlich S, Rothenstein D, Molitoris B, Mazer CD. Teprasiran, a Small Interfering RNA, for the Prevention of Acute Kidney Injury in High-Risk Patients Undergoing Cardiac Surgery: A Randomized Clinical Study. Circulation. 2021 Oct 5;144(14):1133-1144. doi: 10.1161/CIRCULATIONAHA.120.053029. Epub 2021 Sep 3. PMID 34474590